CLINICAL TRIAL: NCT00520481
Title: Phase 2 Single Arm, Open-Label Study of IMC-A12 in Asymptomatic, Chemotherapy-Naïve Patients With Metastatic Androgen-Independent Prostate Cancer
Brief Title: Study With IMC-A12 (Cixutumumab) in Patients Who Have Not Previously Been Treated With Chemotherapy With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 13934; CP13-0603 (Other: ImClone Systems); I5A-IE-JAEJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2007-08-22; First posted 2007-08-24 (Estimated); Results first posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-06

CONDITIONS: Adenocarcinoma of the Prostate
Keywords: prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — cixutumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- IMC-A12 (Experimental): Thirty-one participants will receive IMC-A12 at 10 milligrams per kilogram (mg/kg) administered over 1 hour every other week (every 14 days). An additional 10 participants will receive IMC-A12 at a dose of 20 mg/kg every three weeks. Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met. Radiographic evaluation of response will be performed every 8 weeks for the participants treated with intravenous (i.v.) IMC-A12 at 10 mg/kg and every 9 weeks for the participants treated with i.v. IMC-A12 at 20 mg/kg.
  Interventions: Drug: IMC-A12 (Cixutumumab)

INTERVENTIONS:
Drug: IMC-A12 (Cixutumumab) — 10 mg/kg i.v. infusion over 1 hour every 2 weeks or 20 mg/kg i.v. infusion over 1 hour every 3 weeks.
  Other Names: Cixutumumab; LY3012217

SUMMARY:
This single arm, multicenter, open-label, Phase II study will enroll chemotherapy-naive participants with metastatic, histologically-confirmed adenocarcinoma of the prostate (stage M1 D2). Treatment will continue until there is evidence of disease progression, intolerable toxicity, or other withdrawal criteria are met. Non-surgically castrated participants must continue the use of luteinizing hormone-releasing hormone (LHRH) agonists during protocol treatment.

DETAILED DESCRIPTION:
Thirty-one chemotherapy-naїve participants with asymptomatic metastatic androgen-independent prostate cancer will be enrolled and treated with intravenous (i.v.) IMC-A12 (Cixutumumab) at 10 milligrams per kilogram (mg/kg) administered over 1 hour every 2 weeks. An additional 10 participants will be enrolled and treated with IMC-A12 at a dose of 20 mg/kg every three weeks. Treatment will continue until evidence of disease progression or intolerable toxicity. Radiographic evaluation of response will be performed every 8 weeks for the participants treated with i.v. IMC-A12 at 20 mg/kg.

ELIGIBILITY:
Inclusion Criteria

* The participant is male and at least 18 years of age
* The participant has histologically-confirmed adenocarcinoma of the prostate
* The participant has radiographic evidence of metastatic prostate cancer (stage M1 [D2])
* The participant has prostate cancer unresponsive or refractory to hormone therapy
* The participant must have evidence of progressive disease defined as at least one of the following:

  * a. Progressive measurable disease: using conventional solid tumor criteria.
  * b. Bone scan progression: at least one new lesion on bone scan.
  * c. Increasing prostate specific antigen (PSA): at least two consecutive rising PSA values over a reference value (PSA #1) taken at least 1 week apart. A third PSA (PSA #3) is required to be greater than PSA #2; if not, a fourth PSA (PSA #4) is required to be greater than PSA #2
* The participant has a PSA ≥ 2 nanograms/milliliter (ng/mL)
* The participant has not received prior chemotherapy for metastatic prostate cancer
* The participant had prior surgical or medical castration with a serum testosterone level of < 50 ng/mL. If the method of castration is LHRH agonists, the participant must be willing to continue the use of LHRH agonists during protocol treatment
* All clinically significant toxic effects (excluding alopecia) of prior surgery, radiotherapy, or hormonal therapy have resolved to grade ≤ 1 based on National Cancer Institute - Common Terminology Criteria for Adverse Events, (NCI-CTCAE)Version 3.0
* The participant has not received antiandrogen therapy for at least 6 weeks (4 weeks for flutamide) prior to study entry and is without evidence of an antiandrogen withdrawal response. For participants whose progression is documented solely by PSA increase, the most recent PSA value enabling study entry must be drawn after the required antiandrogen washout period
* The participant has an Eastern Cooperative Oncology Group performance status (ECOG PS) of 0-1
* The participant has adequate organ function including: absolute neutrophil count ≥ 1500/microliter (μL); platelets ≥ 100,000/μL; hemoglobin ≥ 9.0 grams per deciliter (g/dL); bilirubin ≤ 1.5 times the institutional upper limit of normal (ULN); aspartate transaminase (AST) / alanine transaminase (ALT) ≤ 3 times ULN (< 5x ULN if liver metastases are present); creatinine ≤ 1.5 x ULN (or calculated creatinine clearance > 60 milliliter/minute (mL/min); and urine protein ≤ 1+ (if urine protein is ≥ 2+, a 24-hour urine collection must demonstrate < 1000 mg of protein in 24 hours to allow participation in the study)
* The participant has fasting serum glucose < 120 milligrams per deciliter (mg/dL) or below the ULN
* The participant has adequate coagulation function as defined by an international normalized ratio (INR) ≤ 1.5 and a partial thromboplastin time (PTT) ≤ 1.5 ULN (unless on oral anticoagulant therapy). Participants receiving full-dose anticoagulation therapy are eligible provided they meet all other criteria, are on a stable dose of oral anticoagulant or low molecular weight heparin (and if on warfarin have a therapeutic INR between 2 and 3)
* The participant is asymptomatic from prostate cancer. Participants with minimal, infrequent cancer-related symptoms are eligible. Criteria regarding pain and analgesic use are detailed below
* The participant has a life expectancy > 6 months
* The participant, if sexually active, agrees to use contraceptives while on study
* The participant has provided signed informed consent

Exclusion Criteria

* The participant has any active malignancy (other than adequately treated nonmelanomatous skin cancer or other noninvasive or in situ neoplasms), or has an adequately-treated prior cancer but has been disease free for < 3 years
* The participant has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, serious cardiac arrhythmia (well-controlled atrial fibrillation is permitted), psychiatric illness/social situations, active bleeding or pathological condition that carries a high risk of bleeding (eg, tumor involving major vessels, tumor invading to rectal lumen, or known varices), or any other serious uncontrolled medical disorder in the opinion of the investigator
* The participant has a known hypersensitivity to therapeutic protein products
* The participant has known or suspected brain or leptomeningeal metastases
* The participant has received radiotherapy ≤ 21 days prior to first dose of IMC-A12
* The participant has received prior radiation therapy to > 30% of the bone marrow or prior strontium-89, rhenium-186, rhenium-188, or samarium-153 (participants who have received standard dose radiation to the pelvis for prostate cancer and no additional radiotherapy are eligible)
* The participant has a known human immunodeficiency virus infection or acquired immunodeficiency syndrome-related illness
* The participant has received more than one course of radiotherapy to a single site of metastatic bony disease
* The participant has a bone scan that indicates "superscan" (that is (ie), extensive metastasis to bone in numerous areas, too numerous to count or define)
* The participant is receiving corticosteroids (dexamethasone, prednisone, or others) for anorexia, weight loss, analgesia or other cancer-related symptoms(Corticosteroids may not be instituted once a participant has begun therapy on-study
* The participant requires ongoing, regularly scheduled opiate analgesic therapy for cancer related pain. Intermittent, infrequent low-potency opiate-use (example, oxycodone, codeine) is permitted
* The participant has a history of prior treatment with other agents that specifically target the insulin-like growth factor (IGF) receptor

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2007-08; Primary Completion 2012-01 (Actual); Study Completion 2013-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (3):
- United States (3):
  - ImClone Investigational Site, San Francisco, California
  - ImClone Investigational Site, Portland, Oregon
  - ImClone Investigational Site, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Participants who had results for the primary outcome measures were considered to have completed the study. The primary outcome measure is: Composite Time to Disease Progression (cTTP) for Participants Treated With Cixutumumab.
Groups:
- IMC-A12 (Cixutumumab) 10 mg/kg: Cixutumumab was administered at 10 milligrams/kilogram (mg/kg) as intravenous (i.v.) infusion over 1 hour every 2 weeks until disease progression or intolerable toxicity.
- Cixutumumab 20 mg/kg: Cixutumumab was administered at 20 mg/kg as i.v. infusion over 1 hour every 3 weeks until disease progression or intolerable toxicity.
Period: Overall Study
Arm/Group | IMC-A12 (Cixutumumab) 10 mg/kg | Cixutumumab 20 mg/kg
Started | 31 | 10
Received at Least 1 Dose of Study Drug | 31 | 10
Completed | 24 | 9
Not Completed | 7 | 1
Not completed — Adverse Event | 4 | 1
Not completed — Withdrawal by Subject | 3 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug.
Groups:
- Cixutumumab 10 mg/kg: Cixutumumab was administered at 10 mg/kg as i.v. infusion over 1 hour every 2 weeks until disease progression or intolerable toxicity.
- Cixutumumab 20 mg /kg: Cixutumumab was administered at 20 mg/kg as i.v. infusion over 1 hour every 3 weeks until disease progression or intolerable toxicity.
- Total: Total of all reporting groups
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg /kg | Total
Number analyzed (Participants) | 31 | 10 | 41
Age, Continuous [Mean (Standard Deviation); unit: years] | 70.0 (9.26) | 70.2 (6.78) | 70.1 (8.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 31 | 10 | 41
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2
  Not Hispanic or Latino | 29 | 10 | 39
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 10 | 40
  Hispanic | 1 | 0 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 31 | 10 | 41

OUTCOME MEASURES:

1. Primary Outcome: Composite Time to Disease Progression (cTTP) for Participants Treated With Cixutumumab
Description: cTTP was the time from the first day of treatment to the earliest onset of 1 of the following: tumor progression by Response Evaluation Criteria In Solid Tumors [RECIST, version 1.0] criteria: unequivocal evidence of progression by bone scan, new skeletal events, symptomatic progression (for participants without measurable disease), or other clinical events attributable to prostate cancer that in the opinion of the investigator require major interventions. Participants without tumor progression at data cut-off were censored.
Time Frame: From first dose of study drug until progressive disease (Up to 49.2 months)
Population: ITT population: All participants who received at least 1 dose of study drug. Participants censored: Cixutumumab 10 mg/kg =7; or Cixutumumab 20 mg/kg = 2.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Cixutumumab 20 mg/kg: Cixutumumab was administered at or 20 mg/kg as i.v. infusion over 1 hour every 3 weeks until disease progression or intolerable toxicity.
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
months | 4.9 [1.9 to 7.0] | 3.2 [1.0 to 8.8]

2. Primary Outcome: Area Under the Curve (AUC) of IMC-A12 Administered at a Dose of 20 mg/kg Every 3 Weeks
Time Frame: Up to 42 months (predose, 1, 168, 336 and 504 h postdose for Cycles 1 to 4; additionally 24, 72 or 96 h, 120 and 240 or 246 h postdose for Cycle 4; predose and 1 h post dose for Cycles 5 to 9)
Population: Zero participants were analyzed as the data were not estimable accurately due to the study sampling schedule.
Arm/Group | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 0

3. Primary Outcome: Maximum Concentration (Cmax) of IMC-A12 Administered at a Dose of 20 mg/kg Every 3 Weeks
Time Frame: Up to 42 months (predose, 1, 168, 336 and 504 h postdose for Cycles 1 to 4; additionally 24, 72 or 96 h, 120 and 240 or 246 h post dose for Cycle 4; predose and 1 h postdose for Cycles 5 to 9)
Population: Participants who received study drug and had evaluable pharmacokinetic (PK) samples for Cmax on Cycle 1 and Cycle 5.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms/milliliter (µg/ml)
Arm/Group | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 10
micrograms/milliliter (µg/ml)
  After first dose: number analyzed (Participants) | 8
  After first dose | 993 (20)
  After fifth dose: number analyzed (Participants) | 4
  After fifth dose | 1780 (53)

4. Secondary Outcome: Number of Participants Experiencing Serious Adverse Events (SAEs) and Adverse Events (AEs)
Description: Clinically significant events were defined as SAEs and other non-serious adverse events AEs. Participants who died due to progressive disease (PD), AEs while on treatment or died during the 30 day post-treatment are included. A summary of SAEs and other non-serious AEs, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: From randomization up to 49.2 months (and 30 day follow-up)
Population: Safety population: All participants who received any dose of Cixutumumab.
Measure: Count of Participants; unit: Participants
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
Participants
  Non-serious AEs | 28 | 10
  SAEs | 6 | 0
  Deaths due to PD | 1 | 0
  Deaths due to AEs | 1 | 0

5. Secondary Outcome: Time to Radiographically Evident Disease Progression
Description: This is the time between first dose and radiographic progression defined as either: progression of measurable or non measurable lesions using the RECIST v 1.0, evidence of progression by bone scan or new skeletal event including new pathologic bone fracture, new bone lesion requiring radiation or surgery, or spinal cord/nerve root compression. Participants without evidence of disease progression at the date of latest tumor or bone radiograph were censored.
Time Frame: From first dose of study drug until radiographic progression (up to 48.6 months)
Population: ITT population: All participants who received at least 1 dose of study drug. Participants censored: Cixutumumab 10 mg/kg = 9; Cixutumumab 20 mg/kg = 2.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
months | 4.8 [1.9 to 7.5] | 3.3 [1.9 to 8.8]

6. Secondary Outcome: Number of Participants With Complete Response (CR) or Partial Response (PR) (Tumor Response Rate)
Description: Response was defined using RECIST v1.0 criteria: CR was defined as the disappearance of all target lesions and PR was defined as at least a 30% decrease in sum of longest diameter of target lesions
Time Frame: From Randomization up to progressive disease (49.2 months)
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
Participants | 0 | 0

7. Secondary Outcome: Percentage of Participants With Prostate Specific Antigen (PSA) Response Rate
Description: Percentage of participants with a PSA decrease of at least 50% from baseline PSA provided the participant had a PSA value of at least 2 nanograms per milliliter (ng/ml) at baseline. Percentage calculated as: (number of participants with PSA response rate / total number of participants) *100.
Time Frame: From Randomization up to 6.21 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
Participants | 1.0 | 0.0

8. Secondary Outcome: Progression-Free Survival (PFS) Rate at 6 Months
Description: PFS rate was the proportion of participants who had stable disease (SD), PR, or CR and were alive at 6 months after receiving their first dose of study medication. Response was defined using RECIST v1.0 criteria: CR was defined as the disappearance of all target lesions, PR was defined as at least a 30% decrease in sum of longest diameter of target lesions, and SD was defined as shrinkage or increase in tumor size that did not meet the above criteria. For participants not known to have died as of the data cut-off date and who did not have progressive disease, PFS was censored at the date of last visit with adequate assessment. For participants who received subsequent anticancer therapy prior to disease progression or death, PFS was censored at the date of last visit with adequate assessment prior to the initiation of post-discontinuation anticancer therapy. Percentage of participants = (Number of participants with PFS at 6 months / total number of participants analyzed) *100.
Time Frame: From randomization up to 48.6 months
Population: Intent-to-treat (ITT) population: All participants who received at least 1 dose of study drug. Participants censored: Cixutumumab 10 mg/kg - 7; Cixutumumab 20 mg/kg = 2.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Number analyzed (Participants) | 31 | 10
percentage of participants | 41.1 [22.3 to 59.0] | 40.0 [12.3 to 67.0]

9. Secondary Outcome: Area Under the Curve (AUC) of IMC-A12 Administered at a Dose of 10 mg/kg Every 2 Weeks
Time Frame: Up to 42 months (predose and 1 h postdose for Cycles 1, 5, 9, 13, 17 and 21; additionally immediately following dosing, 168 and 336 h postdose for Cycle 1 only)
Population: Zero participants were analyzed as the data were not estimable accurately due to the study sampling schedule.
Arm/Group | Cixutumumab 10 mg/kg
Number analyzed (Participants) | 0

10. Secondary Outcome: Maximum Concentration (Cmax) of IMC-A12 Administered at a Dose of 10 mg/kg Every 2 Weeks
Time Frame: as for outcome 9
Population: Participants who received study drug and had evaluable PK samples for Cmax on Cycle 1 only in 10 mg/kg group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: µg/ml
Arm/Group | Cixutumumab 10 mg/kg
Number analyzed (Participants) | 2
µg/ml | NA (NA) — Per Clinical Study Report, Cmax was not estimated because of small number of participants with evaluable data (n=2). Individual participant data not provided for data privacy reasons.

ADVERSE EVENTS:
Time Frame: From Randomization up to 49.2 months (and 30-day follow-up)
Description: Study-specific clinical outcomes due to progressive disease were not considered to be serious adverse events (SAEs) unless it was deemed related to study drug by the investigator.
Groups:
- Cixutumumab 10 mg/kg: Cixutumumab was administered at 10 mg/kg as intravenous (i.v.) infusion over 1 hour every 2 weeks until disease progression or intolerable toxicity.
- Cixutumumab 20 mg/kg: Cixutumumab was administered at 20mg/kg as i.v. infusion over 1 hour every 3 weeks until disease progression or intolerable toxicity.
Arm/Group | Cixutumumab 10 mg/kg | Cixutumumab 20 mg/kg
Serious Adverse Events (participants affected / at risk) | 6/31 | 0/10
Other Adverse Events (participants affected / at risk) | 28/31 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab 10 mg/kg (N=31) | Cixutumumab 20 mg/kg (N=10)
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 1 (1) | 0 (0)
DISEASE PROGRESSION (General disorders) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 1 (1) | 0 (0)
PNEUMONIA (Infections and infestations) | 1 (1) | 0 (0)
TROPONIN I INCREASED (Investigations) | 1 (1) | 0 (0)
DEHYDRATION (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
FAILURE TO THRIVE (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0)
LEUKOENCEPHALOPATHY (Nervous system disorders) | 1 (1) | 0 (0)
RENAL FAILURE (Renal and urinary disorders) | 2 (2) | 0 (0)
VERTEBRAL ARTERY OCCLUSION (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cixutumumab 10 mg/kg (N=31) | Cixutumumab 20 mg/kg (N=10)
LEUKOCYTOSIS (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 2 (2)
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 (0) | 1 (1)
OEDEMA PERIPHERAL (Cardiac disorders) | 0 (0) | 1 (1)
EAR DISORDER (Ear and labyrinth disorders) | 2 (2) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 2 (2) | 0 (0)
EYELID OEDEMA (Eye disorders) | 0 (0) | 1 (1)
VISUAL DISTURBANCE (Eye disorders) | 5 (7) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 (2) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 5 (5) | 1 (1)
DIARRHOEA (Gastrointestinal disorders) | 5 (5) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 3 (3) | 0 (0)
DYSGEUSIA (Gastrointestinal disorders) | 4 (4) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 11 (15) | 2 (2)
VOMITING (Gastrointestinal disorders) | 5 (7) | 1 (1)
ASTHENIA (General disorders) | 1 (1) | 1 (1)
CHILLS (General disorders) | 0 (0) | 1 (1)
FATIGUE (General disorders) | 12 (20) | 4 (5)
INFUSION RELATED REACTION (General disorders) | 3 (4) | 2 (3)
PYREXIA (General disorders) | 1 (1) | 1 (2)
HYPERSENSITIVITY (Immune system disorders) | 0 (0) | 1 (1)
NAIL INFECTION (Infections and infestations) | 0 (0) | 1 (1)
SINUSITIS (Infections and infestations) | 3 (3) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 4 (5) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (2)
WEIGHT DECREASED (Investigations) | 12 (18) | 2 (3)
ANOREXIA (Metabolism and nutrition disorders) | 5 (5) | 0 (0)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 2 (3) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 6 (9) | 2 (3)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 (9) | 1 (2)
BONE PAIN (Musculoskeletal and connective tissue disorders) | 9 (10) | 2 (5)
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 3 (5) | 0 (0)
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (3)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
MUSCULOSKELETAL DISCOMFORT (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (2)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
SHOULDER PAIN (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
BALANCE DISORDER (Nervous system disorders) | 0 (0) | 1 (1)
DIZZINESS (Nervous system disorders) | 2 (2) | 1 (1)
DYSPHONIA (Nervous system disorders) | 0 (0) | 1 (1)
HEADACHE (Nervous system disorders) | 1 (1) | 1 (1)
HYPOAESTHESIA (Nervous system disorders) | 2 (2) | 0 (0)
INSOMNIA (Nervous system disorders) | 2 (2) | 0 (0)
TREMOR (Nervous system disorders) | 0 (0) | 1 (1)
ANXIETY (Psychiatric disorders) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
PROTEINURIA (Renal and urinary disorders) | 1 (1) | 1 (1)
URINARY INCONTINENCE (Renal and urinary disorders) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
DERMATITIS ALLERGIC (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
ERYTHEMA OF EYELID (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 3 (5) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 3 (4) | 0 (0)
EPISTAXIS (Vascular disorders) | 2 (2) | 0 (0)
HYPOTENSION (Vascular disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Investigators agreed to delay independently publishing or disclosing data, findings or conclusions from the study except as part of a multi-center publication. Upon study publication or if the draft publication is not produced within approximately 6 months of the final report of the study results, investigators may independently publish, subject to confidential information review/redaction by sponsor. The sponsor may request publication delay up to 90 days to seek patent protection.